CLINICAL TRIAL: NCT00481481
Title: A Multicenter, Single-arm, Open, Conversion Study From a Cyclosporine (CyA) Based Immunosuppressive Regimen to a Tacrolimus Modified Release, FK506E (MR4), Based Immunosuppressive Regimen in Kidney Transplant Subjects (CONCERTO: Converting Cyclosporine to FK506E (MR4) in Renal Transplantation)
Brief Title: Conversion Study From Cyclosporine to FK506MR Based Immunosuppression in Kidney Transplant Subjects
Acronym: CONCERTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMR-EC-1209
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Transplantation
Keywords: Tacrolimus, Kidney Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — immunosuppression
  Other Names: Advagraf; FK506MR; MR4

SUMMARY:
Assessment of the safety and the efficacy of a tacrolimus modified release (FK506MR) based immunosuppressive regimen in stable kidney transplant subjects converted from a cyclosporin based immunosuppressive regimen.

DETAILED DESCRIPTION:
Multicenter, single-arm, open phase IIIb, conversion study where a Cyclosporine A-based immunosuppressive regimen is replaced by the administration of tacrolimus modified release formulation, MR4, once daily (morning dosing only) in stable renal transplant subjects. The initial recommended dose of MR4 is 0.1 mg/kg/day.

Twenty-four weeks of treatment on MR4-based immunosuppressive regimen is considered to be an appropriate study duration in order to assess the response in subjects suffering from one or more known cyclosporine side effects, hypertrichosis/hirsutism, gingival hyperplasia, hyperlipidemia, arterial hypertension.

Stable, adult kidney transplant recipients (≥ 12 months post transplant) who are currently treated with cyclosporine and who meet the Inclusion and Exclusion Criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine < 200 µmol/l (< 2.3 mg/dl) at enrollment.
* Female subject of childbearing potential must have a negative serum pregnancy test at enrollment and must agree to maintain effective birth control during the study.
* Capable of understanding the purpose and risks of the study, has been fully informed and has given written informed consent (signed Informed Consent has been obtained).

Exclusion Criteria:

* Previously received an organ transplant other than a kidney.
* Acute rejection episode within 12 weeks prior to enrollment, or an acute rejection episode within the 24 weeks prior to enrollment that required anti-lymphocyte antibody therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in creatinine clearance, calculated according to Cockcroft and Gault formula. | Week 24

SECONDARY OUTCOMES:
Change in creatinine clearance, calculated according to Cockcroft and Gault formula, between Baseline (Day 1) and week 24 (End of Study) overall | Week 24
Rating of subjects according to reason for conversion: Changes in mean lipid levels (total cholesterol) | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma GmbH
Locations (56):
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- Belgium (5):
  - Brussels
  - Edegem
  - Leuven
  - Liège
  - Roeselare
- Czechia (2):
  - Olomouc
  - Prague
- Aarhus, Denmark
- Helsinki, Finland
- France (8):
  - Bordeaux
  - Brest
  - Paris
  - Pierre-Bénite
  - Strasbourg
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Berlin
  - Cologne
  - Essen
  - Halle
  - Hanover
  - Heidelberg
  - Leipzig
  - Lübeck
  - Munich
  - Tübingen
- Hungary (2):
  - Budapest
  - Debrecen
- Italy (11):
  - Bologna
  - Cagliari
  - Florence
  - Genova
  - L’Aquila
  - Milan
  - Modena
  - Napoli
  - Padua
  - Treviso
  - Udine
- Poland (4):
  - Gdansk
  - Lublin
  - Poznan
  - Warsaw
- Spain (7):
  - Alicante
  - Badajoz
  - Barakaldo
  - Madrid
  - Oviedo
  - Palma de Mallorca
  - Salamanca
- Lund, Sweden
- Zurich, Switzerland

REFERENCES:
- [Derived] Rostaing L, Sanchez-Fructuoso A, Franco A, Glyda M, Kuypers DR, Jaray J. Conversion to tacrolimus once-daily from ciclosporin in stable kidney transplant recipients: a multicenter study. Transpl Int. 2012 Apr;25(4):391-400. doi: 10.1111/j.1432-2277.2011.01409.x. Epub 2011 Dec 27. PMID 22211928